CLINICAL TRIAL: NCT03116646
Title: The Reliability and Validity of Family Report Chewing Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, SELEN SEREL ARSLAN, Principal Investigator, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Family report chewing function
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Mastication Disorder
Keywords: mastication; cerebral palsy; family
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chewing evaluation (Experimental): Children with chewing disorders will be recruited. Each child is required to bite and chew a standardized biscuit for chewing evaluation. The chewing function of each child is scored with the Karaduman Chewing Performance Scale by a physical therapist. Then, the chewing function of each child is also scored with the Karaduman Chewing Performance Scale-Family report by their families.
  Interventions: Diagnostic Test: Chewing evaluation

INTERVENTIONS:
Diagnostic Test: Chewing evaluation — Children with chewing disorders will be recruited. Each child is required to bite and chew a standardized biscuit for chewing evaluation. The chewing function of each child is scored with the Karaduman Chewing Performance Scale by a physical therapist. Then, the chewing function of each child is also scored with the Karaduman Chewing Performance Scale-Family report by their families.

SUMMARY:
The family has a primary prescription in the identification of the chewing disorder in children to plan appropriate rehabilitation program and implementation of the training. Therefore, it is very important to investigate the validity and reliability of classification systems that can be applied by parents. The purpose of this study is to determine the validity and reliability of the reliability and validity of family report chewing evaluation.

DETAILED DESCRIPTION:
Chewing is a function that is defined as the grinding of solid food and making them ready for swallowing. Chewing begins with the acceptance of solid food with the lips. The rotational and lateral movements of the tongue is also necessary during grinding the solid food in the molar region. In the molar region, grinding is carried out with the help of salivary and salivary enzymes. Chewing behavior is a learned function. The child begins to chew at 6 months and the coordinated movement to the 9th month continues to develop. Together with experience, chewing activity continues to develop. The families have a primary role in chewing training. In some children, the chewing function does not develop as desired. Many children with developmental, medical, or oral motor problems have difficulty in grinding and swallowing solid foods. Therefore, it is very important to assess the ability of the child's chewing and determine the treatment goals. Assessment of the child's ability to chew should begin by considering chewing as a function. For this reason, the Karaduman Chewing Performance Scale (KCPS) was developed at the Hacettepe University, Faculty of Health Sciences Department of Physiotherapy and Rehabilitation. The chewing performance of the child during chewing a biscuit is scored by the therapist between 0-4. 0 refers to normal chewing, 4 means no bite and chew. The family has a primary prescription in the identification of the chewing disorder in children to plan appropriate rehabilitation program and implementation of the training. Therefore, it is very important to investigate the validity and reliability of classification systems that can be applied by parents. The purpose of this study is to determine the validity and reliability of the reliability and validity of family report chewing evaluation (Karaduman Chewing Performance Scale-Family report).

ELIGIBILITY:
Inclusion Criteria:

* Children above the age of 18 months
* Children with chewing disorders

Exclusion Criteria:

* Children below the age of 18 months
* Children without chewing disorders

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-20 (Actual)

PRIMARY OUTCOMES:
Chewing evaluation | 1 month
  Each child is required to bite and chew a standardized biscuit for chewing evaluation. The chewing function of each child is scored with the Karaduman Chewing Performance Scale.

CONTACTS AND LOCATIONS:
Overall Officials: SELEN SEREL ARSLAN, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacetttepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No